CLINICAL TRIAL: NCT04600869
Title: Effects of Naturalistic Decision-Making Model-based Oncofertility Care Education for Nurses and Patients With Breast Cancer
Brief Title: Effects of Naturalistic Decision-Making Model-based Oncofertility Care Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, the Office of Research and Development, Mackay Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSM/VGH-2017-01-011AC
Record Dates: First submitted 2020-10-16; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Fertility Issues; Breast Cancer; Education
Keywords: Education; Decisional Conflict; Breast Cancer; Nurse; Oncofertility
MeSH Terms: conditions — Infertility; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study examined the effects of an oncofertility education program on decisional conflict in nurses caring for breast cancer patients and patients with breast cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing Group (Experimental): Nurses in the control group accepted the other non-fertility (standard) nursing training for the intervention, whereas those in the experimental group accepted the oncofertility training. Based on research ethics and design, a standard education course was held for the control group after completing data collection in the nursing experimental group. We began to recruit patients into the patient experimental group after all nurses completed their educational courses.
  Interventions: Other: Naturalistic Decision-Making Model-based Oncofertility Care Education

INTERVENTIONS:
Other: Naturalistic Decision-Making Model-based Oncofertility Care Education — We designed the education program according to Klein's NDM model, which explored the reasoning mechanism behind decision-making (Klein, 1993). It depends on the on-the-job training date in each unit. The education program consisted of the following: (1) Information accumulation: explanations of common cancer therapies related to subsequent infertility, psychological and mental change in cancer survivors with infertility, the necessity and method of early determination of fertility intention, and type of fertility preservation. (2) Sense-making: situational case sharing, emphasis on the guidance interaction between experienced and novice nurses to understand the patient's situation. (3) Decision-making: how to provide support, how to correspond, and attitudes toward people with strong fertility intention.

SUMMARY:
his study examined the effects of an oncofertility education program on decisional conflict in nurses caring for breast cancer patients and patients with breast cancer. Other predictors of decisional conflict were also examined.

DETAILED DESCRIPTION:
Background: Nurses play an essential role in transferring knowledge to patients. However, several factors cause nurses to adopt a negative attitude toward providing oncofertility care.

Objective: This study examined the effects of an oncofertility education program on decisional conflict in nurses caring for breast cancer patients and patients with breast cancer. Other predictors of decisional conflict were also examined.

Design: Randomized, controlled experimental research. Settings and Participants: Patients (61) with breast cancer and nurses (79) were recruited from a hospital in Taipei, Taiwan.

Methods: The nursing participants were randomly assigned to receive oncofertility education (experimental group) or usual education (control group). Data from female patients in the control and experimental groups were collected before and after the nurses' educational training, respectively. The oncofertility education consisted of one face-to-face educational session and reading one educational booklet based on the Naturalistic Decision-Making (NDM) Model. The decisional conﬂict was measured using the Chinese version of the decisional conﬂict scale.

ELIGIBILITY:
Inclusion Criteria:

* All nurses involved in breast care were recruited into the study.
* Female patients with breast cancer who were younger than 50 years and who were about to start cancer treatment were recruited from one teaching hospital in Taipei, Taiwan.

Exclusion Criteria:

* Women with a major illness or mental disorder before their cancer diagnosis were excluded.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | Nurses: 1 month; Patients: 6 months
  The decisional conﬂict was measured using the Chinese version of the decisional conﬂict scale. Each item was rated on a five-point Likert scale, ranging from zero to 4. The score was calculated by averaging the sum of individual item scores, then multiplying the product by 25. Hence, the scores range from 0 to 100. A higher score indicates higher decisional conﬂict. Both nursing and patient participants were asked to fill out the questionnaire.
Oncofertility Barrier Scale | Nurses: 1 month
  An Oncofertility Barrier Scale was developed to assess nurses' perceptions of comprehensive barriers regarding oncofertility care. The responses to each item were provided using a five-point Likert scale. A higher scale score meant the nurses perceived that it was more difficult to provide oncofertility care.
Infertility Knowledge Questionnaire | Nurses: 1 month; Patients: 6 months
  We used the Infertility Knowledge Questionnaire to measure both of nurses' and patients' knowledge of infertility in patients with breast cancer. Total scores for the 11 items ranged from zero to 11. Centimeters were used to show the ratio of correct answers visually. A higher score meant a greater level of knowledge about infertility. Both nursing and patient participants were asked to fill out the questionnaire.

SECONDARY OUTCOMES:
Fertility Intention Scale | Patients: 6 months
  The Fertility Intention Scale with 15 items was used to measure patients' fertility intentions. The standardized scale ranged from 1 to 5 points on a five-point Likert scale. Higher scores indicated a greater degree of fertility intention.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Miauh Huang, PhD, Principal Investigator — Department of Nursing, Mackay Medical College
Locations (1):
- Department of Nursing, New Taipei City, Taiwan

REFERENCES:
- [Derived] Huang SM, Tseng LM, Lien PJ. Effects of naturalistic decision-making model-based oncofertility care education for nurses and patients with breast cancer: a cluster randomized controlled trial. Support Care Cancer. 2022 Oct;30(10):8313-8322. doi: 10.1007/s00520-022-07279-w. Epub 2022 Jul 15. PMID 35835904